CLINICAL TRIAL: NCT03681262
Title: Comparing Long-Term Effectiveness of High Frequency and Burst Spinal Cord Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Vafi Salmasi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 47965
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Randomized open label parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High frequency spinal cord stimulation (Experimental): Implant of the device that can deliver high frequency waveform to spinal cord
  Interventions: Device: High frequency spinal cord stimulation
- Burst spinal cord stimulation (Experimental): Implant of the device that can deliver burst waveform to spinal cord
  Interventions: Device: Burst spinal cord stimulation

INTERVENTIONS:
Device: High frequency spinal cord stimulation — We will use Senza® (Nevro Corp., Palo Alto, CA) trial and implant systems to deliver high frequency spinal cord stimulation. A trial system includes two trial leads, an external pulse generator, and a remote control. The permanent implant system includes two leads, an internal pulse generator, a remote control, and a charging device for internal pulse generator. We will use our routine process of trial and implant. High frequency waveform will be delivered with following parameters: frequency of 10,000 hertz, pulse width of 20 microseconds, and amplitude of 0-15 milliamperes.
  Arms: High frequency spinal cord stimulation
Device: Burst spinal cord stimulation — We will use BusrtDRTM (Abbott Saint Jude Medical, St. Paul, MN) trial and implant systems to deliver burst spinal cord stimulation. A trial system includes two trial leads, an external pulse generator, and a remote control. The permanent implant system includes two leads, an internal pulse generator, a remote control, and a charging device for internal pulse generator. We will use our routine process of trial and implant. The parameters of the stimulation are as below: each burst includes 5 pulses of electrical stimulation at intra-burst frequency of 500 hertz without time for discharge in between pulses. These bursts will be repeated at inter-burst frequency of 40-60 hertz. The amplitude will range between 0 and 15 milliamperes.
  Arms: Burst spinal cord stimulation

SUMMARY:
Over 100 million Americans suffer from chronic pain resulting in annual cost of roughly $635 billion. Limited treatments are available for this widespread disease. The data supporting these treatments lack generalizability to patients with more serious medical and psychological comorbidities who are often excluded from explanatory efficacy trials. This study aims to integrate randomized comparative effectiveness research with patient care. The investigators will randomize the patients and collect data using an open-source learning healthcare system already in use in the department to monitor patients' progress: Collaborative Health Outcomes Information Registry (CHOIR). CHOIR uses the National Institute of Health Patient Reported Outcomes Measurement Information System item banks for comparative metrics through computer adaptive testing. The investigators will leverage the advantage of this novel system to compare effectiveness of high frequency and burst spinal cord stimulation in improving pain and function in patients with chronic back and/or leg pain. Spinal cord stimulation is an effective treatment for chronic pain resulting in >50% pain relief in about half of the patients. Novel waveforms for spinal cord stimulation - high frequency and burst - increased the efficacy of this treatment even further. However, there is lack of data guiding decision making of the clinicians in choosing the best waveform in treating the patients with chronic pain. The proposed study will provide the clinicians with this evidence. Currently, data about safety and efficacy of these two novel waveforms is available for up to 24 months. The proposed research will provide data about effectiveness of these two modalities for at least 36 months. Moreover, this study will evaluate feasibility of integrating randomized comparative effectiveness research with patient care in Stanford Pain Management subspecialty clinic. CHOIR can then be applied for numerous future trials to advance knowledge in perioperative and pain medicine.

DETAILED DESCRIPTION:
Specific Aims:

The investigators are proposing to compare the effectiveness of high frequency and burst spinal cord stimulation in patients with chronic back and/or leg pain.

More than one hundred million Americans suffer from chronic pain with estimated annual cost of $635 billion.1 To better characterize these patients, Stanford Pain Management Center has implemented a patient reported registry, Collaborative Health Outcomes Information Registry (CHOIR), since 2012. CHOIR surveys include National Institute of Health (NIH) Patient Reported Outcomes Measurement Information System (PROMIS) item banks, a body map, questions about pain intensity, pain catastrophizing scale, and questions about patients' pain experience and healthcare utilization. This learning healthcare system also has the capability of point-of-care randomization.

Spinal cord stimulation is one of the most effective treatments for patients with intractable trunk and limb pain. Traditional tonic spinal cord stimulation resulted in at least 50% pain reduction in about half of the patients.2,3 Newer waveforms - high frequency and burst - achieve 50% pain reduction in 60-75% of the patients in comparison.4-6 However, more studies are needed to compare effectiveness of these two new waveforms.

The investigators are proposing to use patient reported outcomes to conduct a pragmatic clinical trial that integrates with patients' clinical care; thus, allowing faster recruitment of a larger patient cohort. The patient's provider will use CHOIR point-of-care randomization to randomly assign patients to either receive high frequency or burst spinal cord stimulation. The patients will then complete online CHOIR surveys sent out to them at baseline and then 1, 3, 6, 12, 18, 24 and 36 months after their device implant. These surveys will include PROMIS item banks for pain interference, function, depression and anxiety; questions about pain intensity; and questions about any potential side effects. The investigators will include patients with chronic (pain for at least 6 months) back and/or leg pain refractory to conventional management.

Specific Aim 1: Comparing effectiveness of high frequency and burst spinal cord stimulation in improving pain, function and pain interference in patients with chronic low back and/or leg pain persistent more than 6 months.

The investigators hypothesize that high frequency spinal cord stimulation is more effective than burst spinal cord stimulation in decreasing chronic low back and/or leg pain.

The investigators' primary outcome is change from baseline in pain intensity at 12 months. The investigators will also compare improvement in function and pain interreference at all follow up time points. The investigators will plot the trend of all these measures and study change from baseline at 12 months. The investigators will use repeated measure linear regression to compare these measures between the groups at follow up time points with time as the fixed effect and treatment as random effect.

Specific Aim 2: Comparing effectiveness of high frequency and burst spinal cord stimulation in improving depression and anxiety in patients with chronic low back and/or leg pain persistent more than 6 months.

The investigators hypothesize that high frequency spinal cord stimulation is more effective than burst spinal cord stimulation in decreasing stress and anxiety in patients with chronic low back and/or leg pain.

Burst stimulation modulates medial thalamic pathway, which attributes adverse emotions to pain. The investigators will therefore compare emotional response to these waveforms. The investigators will compare change from baseline of depression and anxiety at 12 months. The investigators will also plot depression and anxiety trend at all follow up time points between two groups using repeated measure linear regression. The investigators will then perform a similar stratified analysis in responders (patients with 50% or more pain reduction at 1 year) and non-responders to these treatments; this analysis is to asses if pain reduction is an effect measure modifier in this relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Adult English-speaking patient 18 years old or above
2. Persistent pain in lower back and/or leg for more than six months
3. Candidate for spinal cord stimulation (with either high frequency or burst waveforms) based on recommendations from Stanford Pain Management Center Neuromodulation Multidisciplinary Team Conference.

Exclusion Criteria:

1. Motor weakness in neurological examination in lower body based on the assessment by treating pain physicians
2. Previous failed spinal cord stimulation trial with either high frequency or burst waveforms
3. Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vafi Salmasi, MD., Principal Investigator — Stanford University
Locations (1):
- Stanford Pain Management Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Frequency Spinal Cord Stimulation: Participants receive a high frequency spinal cord stimulation trial, and receive implant if trial is successful
- Burst Spinal Cord Stimulation: Participants receive a BurstDR spinal cord stimulation trial, and receive implant if trial is successful
Period: Overall Study
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Started | 4 | 3
Received Implant | 4 | 3
Completed Month 12 Survey | 3 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Continuing on study | 3 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >50% Improvement in Pain Intensity
Description: Change from baseline in pain intensity at 12 months. Baseline pain intensity is measured at last CHOIR completion before trial, and is based on patient reported outcome in CHOIR for average pain in the week prior to completion of questionnaire. Score range: 0-10 (higher scores correspond to more severe pain)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Count of Participants; unit: Participants
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
Participants | 2 | 3

2. Secondary Outcome: Number of Participants With Score of 4 or Higher on the Patient Global Impression of Change Survey
Description: Patient global impression of change as Likert scale from 1-5 (higher scores corresponds to more improvement)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Count of Participants; unit: Participants
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
Participants | 2 | 3

3. Secondary Outcome: Pain Intensity Scale Score
Description: Nuremical rating scale of average pain intensity from 0-10 (higher scores corresponds with more severe pain)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
score on a scale | 4.67 (0.47) | 5 (2.94)

4. Secondary Outcome: PROMIS Physical Function T-Score
Description: NIH (National Institute of health) PROMIS (Patient reported outcomes measure information system) function in t-score with population mean of 50 and standard deviation of 10 (higher scores corresponds with worse function)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
t-score | 60.67 (2.05) | 60.33 (4.92)

5. Secondary Outcome: PROMIS Pain Interference T-Score
Description: NIH (National Institute of health) PROMIS (Patient reported outcomes measure information system) pain interference in t-score with population mean of 50 and standard deviation of 10 (higher scores corresponds with worse pain interference)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
t-score | 63 (2.83) | 58.33 (5.25)

6. Secondary Outcome: PROMIS Depression T-Score
Description: NIH (National Institute of health) PROMIS (Patient reported outcomes measure information system) depression in t-score with population mean of 50 and standard deviation of 10 (higher scores corresponds with worse depression)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
t-score | 45 (12.19) | 46 (9.09)

7. Secondary Outcome: PROMIS Anxiety T-Score
Description: NIH (National Institute of health) PROMIS (Patient reported outcomes measure information system) anxiety in t-score with population mean of 50 and standard deviation of 10 (higher scores corresponds with worse anxiety)
Time Frame: 12 months
Population: Participants who completed the surveys
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
Number analyzed (Participants) | 3 | 3
t-score | 48.67 (7.85) | 46.67 (3.3)

ADVERSE EVENTS:
Time Frame: up to 12 months
Arm/Group | High Frequency Spinal Cord Stimulation | Burst Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Frequency Spinal Cord Stimulation (N=4) | Burst Spinal Cord Stimulation (N=3)
Lead Migration (Nervous system disorders) | 1 (1) | 0 — SCS lead migration requiring revision surgery to readjust the leads

LIMITATIONS AND CAVEATS:
Emerging technology halted recruitment, leading to a small number of participants analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03681262/Prot_SAP_000.pdf